CLINICAL TRIAL: NCT01400490
Title: Evaluation of the Biologic Effects of Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA)-Enriched Oils (EPA-DHA Study)
Brief Title: Eicosapentaenoic Acid (EPA)and Docosahexaenoic Acid Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiovascular Research Associates (Network)
Collaborators: Dupont Applied Biosciences (Industry)
Responsible Party: Michael L. Dansinger, MD, Cardiovascular Research Associates
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CVRA 2010-01
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Olive Oil 6 grams/day (Placebo Comparator)
  Interventions: Dietary Supplement: EPA-DHA Study
- DHA 1800 mg/day (Active Comparator)
  Interventions: Dietary Supplement: EPA-DHA Study
- EPA 1800 mg/day (Active Comparator)
  Interventions: Dietary Supplement: EPA-DHA Study
- Fish Oil with EPA 1800 mg/day and DHA 1200 mg/day (Active Comparator)
  Interventions: Dietary Supplement: EPA-DHA Study

INTERVENTIONS:
Dietary Supplement: EPA-DHA Study — 6 weeks of dietary supplementation

SUMMARY:
The goal of the study is to test the efficacy of an EPA-enriched oil made by DuPont versus a DHA-enriched oil, a standard fish oil preparation, and olive oil placebo in a double-blind, randomized, placebo-controlled trial. This study will compare the efficacy of 1800 mg/day of EPA versus 1800 mg/day of DHA versus a fish oil product containing 1800 mg of EPA and 1200 mg of DHA/day as compared to olive oil placebo at 6 grams/day over a 6 week period in a parallel arm design study of 120 healthy adults studied in both the fasting and post-prandial state. Safety will be monitored by assessing for adverse reactions, measuring vital signs and a variety of lab tests including a complete metabolic profile and complete blood count. Efficacy will be assessed by measuring changes in fatty acid profile and or fatty acid ratios,as well as by measuring plasma lipids, lipoproteins, and markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or surgically sterile females between ages 21-70.
* Body Mass Index of 20-35.
* Plasma Lipoprotein Associated Phospholipase A2 (LpPLA2) values > 200 ng/ml.

Exclusion Criteria:

* Competitive exerciser.
* Current smoker.
* Those already taking dietary supplements (EPA, DHA, flax seed oil, fish oil, cod liver oil, weight control products, or high doses of vitamin C (>500 mg/day) or vitamin E (>400 mg/day).
* Those consuming more than 3 oily fish species/week.
* Those consuming >2 drinks containing alcohol/day.
* Those taking medications which could affect serum lipids or body weight, or taking coumadin or more than 325 mg/day of aspirin which could effect bleeding time or the coagulation profile.
* History of a bleeding disorder.
* History of significant cardiac, renal, hepatic, gastro-intestinal, pulmonary, neoplastic, biliary or endocrine disorders including uncontrolled diabetes, thyroid disease, or hypertension.
* Plasma LpPLA2 values < 200 ng/ml.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
plasma EPA levels as well as the EPA/DHA ratio and plasma DHA levels as well as the DHA/EPA ratio | Six weeks
  Subjects receiving EPA at 1800 mg/day will have significantly greater plasma EPA levels as well as the EPA/DHA ratio than the placebo group or the group receiving DHA, while the group receiving DHA will have significantly greater increases in plasma DHA levels as well as the DHA/EPA ratio than the placebo group or the group receiving EPA.

SECONDARY OUTCOMES:
LpPLA2 | 6 weeks
  Subjects receiving the active supplement, especially at the 1800 mg daily dose of EPA will have significant reductions in LpPLA2 as compared to both baseline values and to the placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Research Associates, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tsunoda F, Lamon-Fava S, Asztalos BF, Iyer LK, Richardson K, Schaefer EJ. Effects of oral eicosapentaenoic acid versus docosahexaenoic acid on human peripheral blood mononuclear cell gene expression. Atherosclerosis. 2015 Aug;241(2):400-8. doi: 10.1016/j.atherosclerosis.2015.05.015. Epub 2015 May 19. PMID 26074314